CLINICAL TRIAL: NCT04069767
Title: Innovative Physiotherapy in Stroke Rehabilitation During the Subacute Stage - a Prospective Randomized Single Blinded Controlled Trial and a Qualitative Study
Brief Title: Innovative Physiotherapy in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); Nord University (Other); University of Illinois at Chicago (Other); University of the Basque Country (UPV/EHU) (Other); Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StrokeCoreDIST
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
Keywords: Physiotherapy; Rehabilitation; Trunk Stability; Stroke; Sub-acute; Innovative; Randomized controlled trial; Qualitative study; Gait; Balance
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a parallel trial. After baseline assessment, the participants will be randomly assigned to one of two trial arms, A and B, in a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICoreDIST (Experimental): The intervention starts with an assessment by the physiotherapist to identify the patient's movement problems in order to choose among the 48 exercises in the intervention. Each session lasts for 60 minutes + exercises 5-10 minutes outside of therapy and is performed 5-6 days/per week in the rehabilitation units, and 3 sessions/week + home exercises 30 minutes 3 days per week in home based or outpatient treatment during the 12 weeks period.To allow for individualisation, each exercise contains five levels of difficulty. All exercises demand enhancement of dynamic trunk stability and functional movements.
  Interventions: Procedure: ICoreDIST
- Standard Care (Active Comparator): Consists of standard inpatient rehabilitation, home-based and outpatient-based physiotherapy with the same dose as the intervention group.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Procedure: ICoreDIST — The intervention consists of exercises that demand enhancement of dynamic trunk stability and functional movements, combined with the following:
  1. Optimised alignment and adaptation to the base of support and often using an unstable reference point for the trunk (therapeutic ball) or the distal body parts.
  2. Enhanced somatosensory integration of hands, feet and face, including reduced influence of vision to enhance somatosensory integration.
  3. Proximal stability prior to selective task-oriented movement of limbs, head, eyes.
  4. Inclusion of dual tasks (motor/motor and motor/cognitive) in exercises and activities such as walking indoors, out-doors and climbing stairs.
  5. Specific hands-on interactions or other adaptations to optimise alignment and neuromuscular recruitment.
  6. Exercises combining core activation and moderate increase in heart rate: in lying, sitting, standing and walking.
  Arms: ICoreDIST
Procedure: Standard Care — According to national guidelines for stroke care, every patient in Norway will receive in-patient rehabilitation, home-based and out-patient based physiotherapy.
  Arms: Standard Care

SUMMARY:
The current study has the potential to improve rehabilitation during the subacute phase of a stroke, aiming to reduce the individual's disabilities and risk of falling, enhance health promoting physical activity and independence in ADL.

DETAILED DESCRIPTION:
The purpose of the RCT is to investigate the effects of an innovative physiotherapy intervention, called I-CoreDIST when applied in comprehensive rehabilitation after discharge from a stroke unit and throughout the rehabilitation chain.The project investigate: 1) effects on postural control and balance in various positions and functional activities. Effects on and level of physical activity, and 2) user's identifications of positive and negative features in content and coordination of physiotherapy integrated in post stroke rehabilitation. Function parameters of balance, gait and levels of physical activity at baseline and at 12 weeks will be compared to those obtained from the standard care group. Semistructured interviews will be conducted to identify patients' perceptions of key positive and negative features of content and coordination of I-CoreDIST and standard care rehabilitation after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* A stroke diagnosis
* Can sit for 10 seconds without support
* Age 18-85
* Trunk Impairment Scale-Norwegian version (TIS-NV) < 15
* Pre-stroke modified Ranking Scale (mRS) 0-3

Exclusion Criteria:

* Dementia
* Unable to cooperate in physiotherapy
* On-going substance abuse
* Severe co-morbidity preventing rehabilitation, severe neurological diseases such as Parkinson disease, Multiple Sclerosis and brain tumor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale Norwegian Version | 12 weeks
  Validated scale to assess dynamic sitting balance. The test consists of ordinal 6 sub scales summed to measure dynamic sitting balance and trunk coordination.The scale ranges from 0-16 points where higher score indicates better sitting balance
ActiGraph WgtX-BT | 13 weeks
  Accelerometer recording levels of physical activity and number of steps

SECONDARY OUTCOMES:
Swedish Postural Assessment Scale For Stroke Norwegian Version | 12 weeks
  PASS is a validated postural assessment scale specifically designed to assess and monitor postural control after stroke. It contains 12 four-level items (0-3 points) of varying difficulty for assessing ability to maintain or change a given lying, sitting, or standing posture. The scale ranges from 0-36 points, sub-items are summed to calculate a total score. Higher score indicates better postural control.
MiniBESTest | 12 weeks
  Validated scale to measure pro-and reactive balance in standing and walking
Bodyfitter seat sensor system | 12 weeks
  Pressure mat to register distribution of weight during sitting
Amti Force Platform | 12 weeks
  Device to register postural sway in standing
10 meter walk test | 12 weeks
  Validated test to assess walking speed
2 minute walk test | 12 weeks
  Validated test to assess walking distance
EQ-5D-3L | 12 weeks
  Survey to assess self-perceived quality of life. The EQ-5D-3L comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Stroke Specific Quality of Life Scale | 1 day
  Survey to assess self-perceived quality of life. Stroke-Specific Quality-of-Life (SSQOL) scale is designed to measure multiple effects in poststroke patients. The scale consists of 49 questions grouped into 12 domains. Each domain is assessed on 5-point Gutterman type scales. Provides both summary and domain-specific scores. Domain scores are composed of unweighted averages. Summary scores are composed of an unweighted average of the 12 domain average scores. Scores range from 49-245 and higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Petter Øien, Study Director — Nordlandssykehuset HF
Locations (2):
- Norway (2):
  - Nordlandssykehuset HF, Bodø
  - Sykehuset Levanger, Levanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Normann B, Arntzen EC, Sivertsen M. Comprehensive core stability intervention and coordination of care in acute and subacute stroke rehabilitation-a pilot study. European Journal of Physiotherapy; DOI: 10.1080/21679169.2018.1508497, 2018.
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251